CLINICAL TRIAL: NCT05584995
Title: Uterine Artery Color Doppler Parameters After Bilateral Uterine Artery Ligation for Postpartum Hemorrhage
Brief Title: Uterine Artery Color Doppler Parameters After Bilateral Uterine Artery Ligation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Ossman, Assistant professor, Tanta University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35873/9/22
Record Dates: First submitted 2022-10-11; First posted 2022-10-18 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Postpartum Hemorrhage; Ligation; Color Doppler; Uterine Artery
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): Women will undergo normal cesarean section without Postpartum Hemorrhage or Idiopathic pulmonary hemosiderosis (IPH)
  Interventions: Procedure: Control group
- BUAL group (Experimental): Cases will undergo Bilateral Uterine Artery Ligationafter Postpartum Hemorrhage after cesarean section resistant to medical treatment and did not need a hysterectomy.
  Interventions: Procedure: BUAL group

INTERVENTIONS:
Procedure: Control group — Women will undergo normal cesarean section without Postpartum Hemorrhage or Idiopathic pulmonary hemosiderosis (IPH)
  Arms: Control group
Procedure: BUAL group — Bilateral Uterine Artery Ligation Technique:
  All uterine surgeries will be conducted by externalizing the uterus as much as possible and holding it by the fundus. The BUAL will be done using absorbable suture no. 1 Vicryl (Vicryl 1, Ethicon, France, Neuvilly-sur-Seine, France) will be placed through an avascular space in the broad ligament and tied from the anterior to posterior aspects of the myometrium 2-3 cm medial to the descending portion of the uterine vessels. In all patients, the suture will be carried from the anterior to the posterior at 1 cm to the myometrium medial to the Uterine artery and will be knotted after passing it through the avascular region at 1 cm to the wide ligament section adjacent to the uterus in both sides. All patients will be examined for uterotonics during and after the surgery. The ovarian arteries will be assessed at the level of the ovarian hilum.
  Arms: BUAL group

SUMMARY:
The aim of this study is to assess Uterine artery color doppler parameters after bilateral uterine artery ligation (BUAL) for Postpartum Hemorrhage.

DETAILED DESCRIPTION:
Obstetric haemorrhage is the main reason of maternal death in both countries with high and poor incomes. Most of these deaths occurred within the first 24 hours following birth. Placenta accrete, retained placenta, genital tract lacerations, uterine rupture, and coagulation abnormalities are established risk factors for postpartum hemorrhage. The management of Idiopathic pulmonary hemosiderosis (IPH) and postpartum hemorrhage relies on numerous considerations: type of delivery (vaginal or caesarean delivery), bleeding etiology (uterine atony, trauma, retained placenta) and hemodynamic stability.

In the first stage, early identification, and treatment with uterotonics, suturing the lacerations, and fundal massage are crucial. When bleeding persist, even in the aggressive medical treatment, suitable surgical intervention should be performed.

Surgical therapy relies on the patient's desire to maintain fertility, the severity of the bleeding, and the surgeon's experience.

Historically, peripartum hysterectomy was the only available management to prevent postpartum hemorrhage but, in some instances, hysterectomy alone is insufficient to control the bleeding.

Also, the desire to preserve fertility have resulted in the development of other techniques, such as pelvic embolization and internal iliac artery ligation (IIAL)and bilateral uterine artery ligation (BUAL).

Bilateral uterine artery ligation (BUAL) is the most popular surgical procedure for quick management of postpartum hemorrhage. It may be performed alone or with conjugation with other postpartum hemorrhage methods in with success rate exceeds 90 %. Recanalization is a natural process that may occur following vascular structure closure with a suture or radiological embolization.

ELIGIBILITY:
Inclusion Criteria:

* 70 women aged between 20 and 35 years old.
* Undergoing Bilateral Uterine Artery Ligation after Postpartum Hemorrhageafter cesarean section
* resistant to medical treatment, and did not need to hysterectomy.

Exclusion Criteria:

* Patients with male factor, tubal factor, and absence of lactation.
* Diabetes mellitus, hypertension, morbid obesity, autoimmune disease, or vascular disease in the history, smoking.
* Intrauterine growth restriction in previous pregnancies history, detection of a uterine anomaly or a medical condition, as well as administration of a hormonal treatment during the study.
* Uncontrolled bleeding is needed for a hysterectomy.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 70 women aged between 20 and 35 years old. Cases underwent Bilateral Uterine Artery Ligation after Postpartum Hemorrhageafter cesarean section, resistant to medical treatment, and did not need to hysterectomy. The Control group will undergo normal cesarean section without Postpartum Hemorrhage or Idiopathic pulmonary hemosiderosis (IPH)
Enrollment: 70 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Color Doppler parameters | After Bilateral Uterine Artery Ligation
  Color Doppler parameters for measuring the UtA diameters as UtA pulsatility Index will be recorded

SECONDARY OUTCOMES:
The uterine artery's descending branches | After Bilateral Uterine Artery Ligation
  The uterine artery's descending branches will be measured at the level of the internal os of the uterine cervix.
The uterine artery's ascending branch | After Bilateral Uterine Artery Ligation
  The uterine artery's ascending branch on the left and right sides of the uterine isthmus will be identified by means of color flow imaging to obtain uterine arterial blood flow velocity waveforms.
Color Doppler parameters | After Bilateral Uterine Artery Ligation
  resistance Index (RI) will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed M.E. Ossman, Tanta, El-Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available under a reasonable request from the corresponding author.
Supporting Information: Study Protocol
Time Frame: One year after the end of the study